CLINICAL TRIAL: NCT07340255
Title: The 90% Effective Ventilation Pressure (EP90) for Esophageal Insufflation Avoidance During Anesthesia Induction: A Bias-Coin Design With Up-and-Down Sequential Allocation Trial
Brief Title: The 90% Effective Ventilation Pressure (EP90) for Esophageal Insufflation Avoidance During Anesthesia Induction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Jiaxing University (Other)
Responsible Party: Principal Investigator, Qing-he Zhou, Director, Head of Anesthesiology, Affiliated Hospital of Jiaxing University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-KY-396
Record Dates: First submitted 2025-09-28; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Airway Management; Induction of Anesthesia
Keywords: Esophageal Insufflation; Airway Management; Ventilation; Bias-coin Design
MeSH Terms: conditions — Respiratory Aspiration | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ventilation Pressure (Experimental): Anesthesia machine settings: pressure control mode, inspiratory-to-expiratory ratio of 1:2, respiratory rate of 15 breaths/min, 100% oxygen, no PEEP applied. Mask ventilation duration was standardized to 120 seconds, followed by tracheal intubation.
  Interventions: Other: Ultrasonic and inflation determination

INTERVENTIONS:
Other: Ultrasonic and inflation determination — Before induction, during ventilation, and after intubation, the anesthesiologist used a 7-14 MHz linear array probe for transverse (supraclavicular) positioning to monitor the left paratracheal esophageal region in real time. The main criterion for assessment was the absence of esophageal gas during ventilation, which was considered a positive response. If gas was detected entering the esophagus on ultrasound, it was recorded as a negative response.
  Additionally, the anesthesiologist performed a preoperative ultrasound examination of the gastric antrum to record baseline gastric antrum parameters. After successful tracheal intubation, a follow-up ultrasound of the gastric antrum was conducted to obtain postoperative gastric antrum parameters.

SUMMARY:
Exploring the 90% Effective Ventilation Pressure (EP90) for Esophageal Insufflation Avoidance During Anesthesia Induction: The aim is to determine the optimal ventilation pressure for esophageal insufflation avoidance during anesthesia induction and to explore its guiding significance for anesthesia management. The goal is to provide a more precise and personalized ventilation pressure setting standard for clinical anesthesia, thereby enhancing the safety of the anesthesia induction phase.

DETAILED DESCRIPTION:
Pulmonary aspiration of gastric contents has been identified as one of the leading causes of anesthesia-related mortality. Even in fasting patients or those without known aspiration risks, such complications can still occur. In fact, in patients with unprotected airways during apnea, the introduction of air into the lungs during ventilation may become a potential trigger for gastric content aspiration. The entry of air can increase gastric pressure, leading to the reflux of gastric contents into the esophagus, which may subsequently result in hemodynamic instability and pulmonary failure. Therefore, airway management during anesthesia induction is crucial, particularly in the precise control of ventilation pressure, as it directly impacts the safety of the patient during surgery.

Previous studies have used gastric insufflation as the primary endpoint for evaluating the safety of ventilation pressures, often assessing the appearance of gastric gas in the stomach during mask ventilation. However, gastric insufflation typically occurs only after gas has passed through the esophagus and cardia, entering the gastric cavity-this process is a "terminal event" triggered by higher pressures. The esophagus, being structurally weaker than the stomach, is less tolerant to pressure. When gas first enters the esophagus, the cardia is not fully open, and if ventilation pressure continues to rise, it is easy to cause esophageal insufflation, further leading to gastric insufflation and even gastric content reflux. Since esophageal insufflation occurs earlier and has a lower pressure threshold, it can serve as a more sensitive indicator, providing an early warning to anesthesiologists about potential airway management issues.

To address this issue, determining the optimal ventilation pressure to avoid esophageal insufflation is particularly important. the 90% effective ventilation pressure (EP90) refers to the ventilation pressure that can avoid esophageal insufflation in 90% of cases, providing anesthesiologists with a quantitative reference for ventilation pressures.

This study employed a Sequential Allocation with Biased Coin Design (SABCD) trial, utilizing precise statistical methods to explore the EP90 for avoiding esophageal insufflation during anesthesia induction. The goal was to determine the optimal ventilation pressure for preventing esophageal insufflation during anesthesia induction and to explore its implications for anesthesia management. The ultimate aim is to provide a more precise and personalized ventilation pressure setting standard for clinical anesthesia, thereby enhancing the safety of the anesthesia induction phase.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65 years, regardless of gender;
2. ASA classification: I-III;
3. Scheduled for elective general anesthesia surgery;
4. BMI: 18.0-28.0 kg/m²;
5. Preoperative fasting: Solid food >6 hours, liquid >2 hours;
6. Less than two from five criteria predicting difficult mask ventilation as described by Langeron et al.(Prediction of difficult mask ventilation. Anesthesiology 2000; 92:1229-36);
7. No severe underlying conditions such as heart, lung, liver, or kidney disease;
8. Signed informed consent and ability to cooperate with the study protocol.

Exclusion Criteria:

1. Pregnant or breastfeeding women;
2. History of upper gastrointestinal diseases such as gastroesophageal reflux disease, peptic ulcers, or hiatal hernia;
3. Recent (within 2 weeks) respiratory infections, chronic cough, similar symptoms, and other known or predictable respiratory system diseases;
4. Need for emergency surgery or airway obstruction after anesthesia induction requiring urgent intubation;
5. Inability to achieve adequate oxygenation during mask ventilation (e.g., SpO₂ < 92% for 30 seconds, unresponsive to treatment);
6. History of contraindications or allergies to study medications;
7. Inability to understand the study content or refusal to cooperate;
8. Oropharyngeal or facial pathology;
9. with an indwelling gastric tube, and who had previously undergone gastric surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
EP90 | Perioperative
  The 90% effective ventilation pressure (EP90) for avoiding esophageal inflation refers to the minimum effective airway pressure (measured in cmH₂O) at which 90% of patients do not experience esophageal inflation during pressure-controlled mask ventilation during anesthesia induction.

SECONDARY OUTCOMES:
EP95 | Periprocedural
  The 95% effective ventilation pressure (EP95) for avoiding esophageal inflation refers to the minimum effective airway pressure (measured in cmH₂O) at which 95% of patients do not experience esophageal inflation during pressure-controlled mask ventilation during anesthesia induction.
EP98 | Periprocedural
  The 98% effective ventilation pressure(EP98) for avoiding esophageal inflation refers to the minimum effective airway pressure (measured in cmH₂O) at which 98% of patients do not experience esophageal inflation during pressure-controlled mask ventilation during anesthesia induction.
Ventilation-related respiratory parameters | Periprocedural
  pulse oxygen saturation (SpO₂) was recorded at multiple time points during mask ventilation and 30/60/90/120 seconds after tracheal intubation.
Ventilation-related respiratory parameters | Periprocedural
  end-tidal carbon dioxide (EtCO₂) was recorded at multiple time points during mask ventilation and 30/60/90/120 seconds after tracheal intubation.
Ventilation-related respiratory parameters | Periprocedural
  end-tidal oxygen concentration (EtO₂) was recorded at multiple time points during mask ventilation and 30/60/90/120 seconds after tracheal intubation.
Ventilation-related respiratory parameters | Periprocedural
  minute leak volume was recorded at multiple time points during mask ventilation and 30/60/90/120 seconds after tracheal intubation.
Ventilation-related respiratory parameters | Periprocedural
  peak airway pressure (Ppeak) was recorded at multiple time points during mask ventilation and 30/60/90/120 seconds after tracheal intubation.
Ventilation-related respiratory parameters | Periprocedural
  tidal volume (Vt) was recorded at multiple time points during mask ventilation and 30/60/90/120 seconds after tracheal intubation.
Incidence of complications Incidence of complications | Periprocedural
  Including gastric distension, signs of aspiration, failure rate of mask ventilation [such as pulse oxygen saturation (SpO₂) < 92% lasting for 30 seconds], intubation condition score (Cormack-Lehane classification), hypoxemia and other adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Qinghe Zhou, Dr., Study Chair — Affiliated Hospital of Jiaxing University
Locations (1):
- Affiliated Hospital of Jiaxing University, Jiaxing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Langeron O, Masso E, Huraux C, Guggiari M, Bianchi A, Coriat P, Riou B. Prediction of difficult mask ventilation. Anesthesiology. 2000 May;92(5):1229-36. doi: 10.1097/00000542-200005000-00009. PMID 10781266